CLINICAL TRIAL: NCT03148223
Title: Effect of Auriculotherapy in the Treatment of Dysmenorrhea: Protocol of a Randomized Controlled Clinical Trial
Brief Title: Auriculotherapy in the Treatment of Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sorocaba (Other)
Responsible Party: Principal Investigator, Luciane Cruz Lopes, Responsible researcher, University of Sorocaba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 45269015.3.0000.5500
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; acupuncture; auriculotherapy
MeSH Terms: conditions — Dysmenorrhea | interventions — Auriculotherapy; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be informed which group they belong to, intervention or control. Who will apply the treatment will not be blind, since during the treatment it will know if the points to be stimulated must contain seeds of mustard or just plaster, but will not have previous knowledge of the members of the groups. The evaluator, who is responsible for applying the pre- and post-treatment evaluation instruments, will be blind and not aware of the research intervention. The data analyst will also be early for the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Auriculotherapy with application of mustard seeds fixed with adhesive tape at specific points in the auricle during one session per week lasting 20 minutes for 3 consecutive months.
  Interventions: Device: auriculotherapy
- Control (Placebo Comparator): Auriculotherapy with tape-only fixation in the auricle, without mustard seeds, following the same stitch protocol used with the intervention group, during a session per week lasting 20 minutes, for three consecutive months.
  Interventions: Device: auriculotherapy

INTERVENTIONS:
Device: auriculotherapy — The participants will be submitted to a session per week with duration of 20 minutes, for three consecutive months, to fix the adhesives. The points selected for stimulation, according to Chinese atrial mapping, are: uterus, endocrine, ovary, pituitary, shen men, sympathetic, and liver. Participants will be advised to remain with the stickers fixed to the auricle for six days.
  Other Names: acupuncture

SUMMARY:
This study aims to determine if auriculotherapy is effective in the treatment of dysmenorrhoea. This intervention consists of fixation of yellow mustard seeds at specific points of the auricular pavilion (or area), with opaque tape. Half of the participants will have specific ear pinch points stimulated by mustard seeds fixed with opaque plaster, while the other half will have only the adhesive plasters fixed, without the seeds for stimulation.

DETAILED DESCRIPTION:
Primary dysmenorrhoea is responsible for the most part of dissatisfactions in the female class, in the face of discomforts which are caused monthly. For this, the income index of this woman in the work environment tends to reduce, thus harming the development of every sector to which she responds. The expected effects, after the intervention, will be positive, favoring a considerable improvement of the symptoms reported by the women. We chose auriculotherapy because it is a non-medicated, noninvasive intervention that is inexpensive.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, the individual must meet the following criteria:

  * Free and informed consent form, duly signed and dated
  * Consent to voluntarily participate in all study procedures and availability for the duration of the study
  * Female subjects
  * Age above of 18 years old
  * Enjoy good general health
  * Have active menstrual cycle
  * Complaint about dysmenorrhea

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * Clinical diagnosis of endometriosis
  * Myomas
  * Pelvic inflammatory disease
  * Adenomyosis
  * In the active phase for treatment of cancer (chemotherapy or radiotherapy)
  * Women who are already in menopause
  * Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Measurement on pain perception | 12 weeks
  The numerical visual scale of pain 0-10 (0 = no pain, 10 = worst possible pain), applied at the beginning of the intervention period and reapplied to each menstrual period during the 12 weeks of follow-up will be used.

SECONDARY OUTCOMES:
Welfare | 12 weeks
  The quality of life questionnaire (Short-Form Health Survey SF36) will be applied at the beginning of the intervention period and reapplied at the end of the 12 weeks of intervention.
Number of participants with adverse events | 12 weeks
  Adverse events will be collected spontaneously by the active survey, at all visits of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Luciane Cruz Lopes, Principal Investigator — Universidade de Sorocaba
Locations (1):
- Universidade de Sorocaba - Campus Cidade Universitária, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We intend to share the data six months after the conclusion of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available since the study were published.
Access Criteria: Data access requests should be made via an application form detailing the specific requirements and the proposed research and publication plan. Any request access will be controlled to types of data analyses, process for requesting data/documents. We will discuss with the team of researcher the "quality of request".
URL: http://www.uniso.br

REFERENCES:
- [Background] Chan AW, Hrobjartsson A, Haahr MT, Gotzsche PC, Altman DG. Empirical evidence for selective reporting of outcomes in randomized trials: comparison of protocols to published articles. JAMA. 2004 May 26;291(20):2457-65. doi: 10.1001/jama.291.20.2457. PMID 15161896
- [Background] Dawood MY. Primary dysmenorrhea: advances in pathogenesis and management. Obstet Gynecol. 2006 Aug;108(2):428-41. doi: 10.1097/01.AOG.0000230214.26638.0c. PMID 16880317
- [Background] Latthe P, Latthe M, Say L, Gulmezoglu M, Khan KS. WHO systematic review of prevalence of chronic pelvic pain: a neglected reproductive health morbidity. BMC Public Health. 2006 Jul 6;6:177. doi: 10.1186/1471-2458-6-177. PMID 16824213
- [Background] Weissman AM, Hartz AJ, Hansen MD, Johnson SR. The natural history of primary dysmenorrhoea: a longitudinal study. BJOG. 2004 Apr;111(4):345-52. doi: 10.1111/j.1471-0528.2004.00090.x. PMID 15008771
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Background] Altman DG, Bland JM. How to randomise. BMJ. 1999 Sep 11;319(7211):703-4. doi: 10.1136/bmj.319.7211.703. No abstract available. PMID 10480833
- [Background] Smith CA, Armour M, Zhu X, Li X, Lu ZY, Song J. Acupuncture for dysmenorrhoea. Cochrane Database Syst Rev. 2016 Apr 18;4(4):CD007854. doi: 10.1002/14651858.CD007854.pub3. PMID 27087494
- [Background] Song JS, Liu YQ, Liu CZ, Xie JP, Ma LX, Wang LP, Zheng YY, Ma ZB, Yang H, Chen X, Shi GX, Li SL, Zhao JP, Han JX, Wang YX, Liu JP, Zhu J. [Cumulative analgesic effects of EA stimulation of sanyinjiao (SP 6) in primary dysmenorrhea patients: a multicenter randomized controlled clinical trial]. Zhen Ci Yan Jiu. 2013 Oct;38(5):393-8. Chinese. PMID 24308187